CLINICAL TRIAL: NCT04585399
Title: Increasing MAT Engagement With Contingency Management Among Individuals With Opioid Use Disorder in an ED Bridge Program
Brief Title: Increasing MAT Engagement With Financial Incentives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Collaborators: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-112EX
Record Dates: First submitted 2020-03-09; First posted 2020-10-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Two group, randomized controlled trial.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Participants will only told if they are assigned to the contingency management group because there are different procedures for those individuals. The care providers will not know which participants are in the control group but they may know when people are in the CM group because extra urine screens will be collected and they will be scheduled for rides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contingency Management (Experimental): Participants in this arm of the study will receive financial incentives for attending their buprenorphine appointments and for being clean from other opioids. Participants in this group will also have up to two rides per week paid for to attend bup appointments.
  Interventions: Behavioral: Contingency management
- Standard Care (No Intervention): Participants in this group will be treatment as usual and will not receive any incentives for attending their bup appointments or for being opioid abstinent.

INTERVENTIONS:
Behavioral: Contingency management — Financial incentives for attending bup appointments and demonstrating opioid abstinence. Rides will also be provided for up to two clinic visits per week.
  Arms: Contingency Management

SUMMARY:
The increased prevalence of opioid use disorder (OUD) and associated overdoses and adverse events has led to a substantial increase in the number of patients being seen at emergency departments (ED). Thus, the ED may be an ideal location for identifying patients in need of OUD treatment and can serve as the first touch point in the OUD continuum of care to promote medication assisted treatment initiation. Contingency management (CM) is an effective method for promoting treatment initiation and adherence that has not been thoroughly evaluated for this purpose. The primary aim of the current study is to develop and assess the effectiveness, acceptability, and feasibility of a protocol for delivering CM to increase combined buprenorphine + nalaxone (referred to as BUP hereafter) initiation and continuous adherence for OUD in an existing ED "bridge" program (e.g., Bridge plus CM; B+CM) relative to standard care. Secondary objectives include identifying behavioral and neuropsychological correlates to treatment outcomes, including delay discounting, reinforcer demand, and neurological soft signs.

ELIGIBILITY:
Inclusion Criteria:

1. Participants at least 18 years of age
2. Participants must be newly enrolled in the Bridge program in the Cooper University ED, with their first clinic appointment scheduled to take place at the Cooper Outreach Clinic within one week of enrollment.
3. All subjects must be in good physical health as determined by a physical examination and premenopausal women will have a pregnancy test on the day of the study to rule out pregnancy

Exclusion Criteria:

1. Participants who demonstrate contraindication with Suboxone treatment or who are currently or have recently used other medication-assisted therapies for opioid use disorder.
2. Participants who are currently pregnant or breastfeeding or have been diagnosed with a DSM-5 psychiatric condition that might interfere with treatment delivery (e.g., uncontrolled schizophrenia, bipolar disorder, dementia)
3. Participants who are non-English speaking or cannot otherwise provide valid informed consent.
4. Individuals who are unable to complete the survey assessments, due to literacy or visual impairments.
5. The participant will not be a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Attendance at first scheduled clinic appointment | 1 week
  We will track attendance at participant's first scheduled BUP appointment after being bridged from the ED
Percentage of sessions where buprenorphine positive urine results was recorded | 3-months
  Urine-verified buprenorphine
Percentage of sessions where opioid free urine results were recorded | 3-months
  Urine-verified opioid abstinence
Treatment acceptability | 3-months
  Participants will evaluate the treatment at the end.

SECONDARY OUTCOMES:
Delay discounting as a correlate of opioid-free urine test results and buprenorphine-positive results | 3-months
  Delay discounting will be evaluated, using the brief, five question delay discounting procedure and will be correlated with urine results determining opioid abstinence and buprenorphine adherence.
Opioid demand as a correlate of opioid-free urine test results and buprenorphine-positive results | 3-months
  The opioid purchasing task will be used to evaluate opioid demand and will be correlated with urine results determining opioid abstinence and buprenorphine adherence.
Substance-free activities as a correlate of opioid-free urine test results and buprenorphine-positive results | 3-months
  A modified Pleasant Events Scale survey will be used to evaluate access to, and enjoyment from, substance-free activities and the results will be correlated with urine results determining opioid abstinence and buprenorphine adherence.
Neurological Soft Signs correlate with treatment success | 3-months
  Participants will complete a drawing task that has been correlated with other substance use treatment outcomes in the past.

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will share the data after we have completed the study and have published all of the outcomes. We will only share the data with qualified researchers who provide a written request with clear justification for their need to access the data.

REFERENCES:
- [Derived] Goodwin SR, Kirby KC, Salzman MS, Raiff BR. Pragmatic and low-cost contingency management intervention increases buprenorphine treatment engagement: Randomized controlled trial. Exp Clin Psychopharmacol. 2026 Feb;34(1):68-77. doi: 10.1037/pha0000823. PMID 41538228